CLINICAL TRIAL: NCT03239548
Title: "A Study to Assess the Opinion of Doctors, Nurses and Key Informants Regarding Independent Nurse Midwifery Practitioner at Selected Hospitals and Colleges of Nursing in Haryana."
Brief Title: "Opinion of Doctors,Nurses and Key Informants About Independent Nurse Midwifery Practitioner in Northern India
Acronym: INMP
Status: Completed | Type: Observational
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Shikha Guleria, Principal Investigator, Maharishi Markendeswar University (Deemed to be University)
Other Study IDs: 100076
Record Dates: First submitted 2017-08-01; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Opinion
Keywords: Opinion,; Doctors,; Nurses,; Key informants,; Independent Nurse Midwifery Practitioner

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Doctor: It refers to the doctors with minimum qualification as M.B.B.S and B.A.M.S; working on various posts in the clinical areas of all the departments of selected hospitals.
- Nurses: It refers to the Registered Nurses working on various posts in the clinical areas of all the departments of selected hospitals and Principals, Vice Principals of selected colleges.
- Key informants: It refers to the general public including patients admitted and attending O.P.D and their attendants with minimum qualification as graduation.

SUMMARY:
"A Study to assess the Opinion of Doctors, Nurses and Key informants regarding Independent Nurse Midwifery Practitioner at selected Hospitals and Colleges of nursing in Haryana."

DETAILED DESCRIPTION:
Abstact Introduction: Despite improvement in coverage of institutional deliveries and skilled birth attendants, India has missed its Millennium Development Goal to reduce maternal mortality rate. In order to increase access to primary care services, the Independent Nurse Practitioner (INP) is one of the best solutions.

Objectives: The objectives of the study were to assess the opinion of doctors, nurses and key informants regarding Independent Nurse Midwifery Practitioner (INMP) and to determine the association of opinion score of doctors, nurses and key informants with their selected demographic variables.

Material and Methods: A Quantitative Non Experimental Research Approach and Descriptive Survey Design was adopted. A total of 400 subjects (120 doctors, 120 nurses and 160 key informants) were selected using purposive sampling technique from selected hospitals and nursing colleges of Ambala, Panchkula and Yamunanagar districts of Haryana. The tool used for the study consisted of structured performa regarding sample characteristics and likert scale. Research tool was submitted to 11 experts from various departments for validity. Reliability was calculated by Cronbach's alpha and it was 0.75 for likert scale. Data Collection was done from December 2016 to February 2017. The obtained data was analyzed and interpreted in terms of objectives and research hypothesis. Descriptive and inferential statistics were used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Doctors, nurses and key informants who were

  * available at the time of data collection in study setting.
  * willing to participate in the study.
  * able to read and write Hindi or English.

Exclusion Criteria:

* Key informants who were not having minimum qualification as graduation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Doctors, nurses and key informants in selected hospitals and colleges of Panchkula, Ambala and Yamunanagar districts of Haryana and available during data collection.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Likert scale | 12-15 Minutes
  A Structured likert scale was developed to assess the opinion of doctors, nurses and key informants regarding Independent Nurse Midwifery Practitioner. Likert scale consisted of 26 items prepared to assess the opinion of doctors , nurses and key informants regarding Independent Nurse, Midwifery Practitioner.
  It consists of 13 positive items and 13 negative items.The respondent was required to give their opinion on likert's five point scale from strongly agree, agree, undecided, disagree and strongly disagree. The responses were quantified by giving scores. Every positive statement was scored as:Strongly agree - 5, Agree - 4, Undecided - 3, Disagree - 2 and Strongly disagree - 1. And every negative statement was scored as:Strongly agree - 1, Agree - 2, Undecided - 3, Disagree - 4 and Strongly disagree - 5. The maximum score was 130 and minimum score was 26. It consists score of 98 -130 (Favourable), 65 - 97 (Moderately favorable) and 26 - 64 (Unfavouable)

CONTACTS AND LOCATIONS:
Overall Officials: Poonam Sheoran, Ph.D Nursing, Study Director — Maharishi Markandeshwar University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoll KH, Hauck YL, Hall WA. Home or hospital? Midwife or physician? Preferences for maternity care provider and place of birth among Western Australian students. Women Birth. 2016 Feb;29(1):e33-8. doi: 10.1016/j.wombi.2015.07.187. Epub 2015 Aug 28. PMID 26319505